CLINICAL TRIAL: NCT03591393
Title: Pelvic Floor Dysfunction and Its Influence on Body Image and Sexual Function - A Prospective Study Through Pregnancy and Post-partum
Brief Title: Pelvic Floor Dysfunction and Its Influence on Body Image and Sexual Function
Acronym: PFD-BI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S60939
Record Dates: First submitted 2018-06-05; First posted 2018-07-19 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Body Image; Urinary Incontinence; Anal Incontinence; Anorectal Disorder; Constipation; Pelvic Organ Prolapse; Sexual Dysfunction; Pregnancy Related; Postpartum Disorder
MeSH Terms: conditions — Urinary Incontinence; Encopresis; Rectal Diseases; Constipation; Pelvic Organ Prolapse; Sexual Dysfunction, Physiological; Puerperal Disorders | interventions — Pain Measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant women (Experimental): * questionnaire at 1st and 3rd trimester, 10-12 weeks postpartum and 12 months postpartum
  * pelvic floor ultrasound at 1st trimester and at 3rd trimester
  Interventions: Diagnostic Test: questionnaire

INTERVENTIONS:
Diagnostic Test: questionnaire — Validated self-administered questionnaires with five domains: Wexner questionnaire for anal incontinence, PAC-SYM for constipation, International Consultation on Incontinence Questionnaire Short Form for urinary incontinence, the Pelvic Organ Prolapse Distress Inventory for pelvic organ prolapse, POP/UI Sexual Questionnaire - IUGA revised for sexual function.
  The body image perception will be assessed using the Dutch-validated version of the self-administered Body Image Disturbance Questionnaire.
  Other Names: pelvic floor ultrasound

SUMMARY:
The first objective to determinate the prevalence of pelvic floor dysfunction in pregnant women and in the first year postpartum. The second objective is to assess the anatomical (both clinical and ultrasound), demographic and obstetric variables in symptomatic women and their association with pelvic floor dysfunction, sexual function and Body Image.

This is a single center prospective cohort study. Women will be asked to fill out a questionnaire at the time of their 1st and 3rd trimester scan, at the postpartum checkup and 12 months postpartum. Furthermore, they will undergo a pelvic floor ultrasound at the time of their first and third trimester scan.

The presence of pelvic floor dysfunctions will be recorded through validated self-administered questionnaires with five domains: Wexner questionnaire for anal incontinence, PAC-SYM for constipation, International Consultation on Incontinence Questionnaire Short Form for urinary incontinence, the Pelvic Organ Prolapse Distress Inventory for pelvic organ prolapse, POP/UI Sexual Questionnaire - IUGA revised for sexual function.

The body image perception will be assessed using the Dutch-validated version of the self-administered Body Image Disturbance Questionnaire.

The anatomy of the pelvic floor will be objectively assessed off line on 3D/4D transperineal ultrasound volumes and POP-Q examination. The demographic variables and information about the pregnancy and the delivery will be obtained from the medical records.

ELIGIBILITY:
Inclusion Criteria:

* age > or = 18 years
* dutch-speaking
* ongoing pregnancy before 14 weeks GA
* intending to deliver in UZ Leuven
* ICF

Exclusion Criteria:

* age < 18 years
* not dutch-speaking
* non evolutive pregnancy
* pregnancy over 14 weeks GA
* intention to deliver elsewhere

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Change Body Image during and after pregnancy | through study completion, an average of 18 months
  Body Image Disturbance Questionnaire Score: 7-item questionnaire, each item is scored on a 5-point Likert-scale (1=no disturbance at all; 5=extreme disturbance), the final score is the mean of the 7-item ordinal scores.

SECONDARY OUTCOMES:
Urethra mobility in cm | 11-13 weeks gestation
  Transperineal ultrasound
Urethra mobility in cm | 28-33 weeks gestation
  Transperineal ultrasound
genital hiatus in cm^2 | 11-13 weeks gestation
  Transperineal ultrasound
genital hiatus in cm^2 | 28-33 weeks gestation
  Transperineal ultrasound
levator ani avulsion | 11-13 weeks gestation
  TUI sequence
levator ani avulsion | 28-33 weeks gestation
  TUI sequence
anal sphincter injury | 11-13 weeks gestation
  TUI sequence
anal sphincter injury | 28-33 weeks gestation
  TUI sequence
Urinary Incontinence | 11-13 weeks gestation
  International Consultation Incontinence Questionnaire - short form
Urinary Incontinence | 28-33 weeks gestation
  International Consultation Incontinence Questionnaire - short form
Urinary Incontinence | 3 months postpartum
  International Consultation Incontinence Questionnaire - short form
Urinary Incontinence | 12 months postpartum
  International Consultation Incontinence Questionnaire - short form
Anal Incontinence | 11-13 weeks gestation
  wexner score: 5-items questionnaire measuring the frequency of complaints. Each item is scored 0-4 (0=never, 4=always). The final score is the sum of the scores of the 5 items (total score 0-20)
Anal Incontinence | 28-33 weeks gestation
  wexner score: 5-items questionnaire measuring the frequency of complaints. Each item is scored 0-4 (0=never, 4=always). The final score is the sum of the scores of the 5 items (total score 0-20)
Anal Incontinence | 3 months postpartum
  wexner score: 5-items questionnaire measuring the frequency of complaints. Each item is scored 0-4 (0=never, 4=always). The final score is the sum of the scores of the 5 items (total score 0-20)
Anal Incontinence | 12 months postpartum
  wexner score: 5-items questionnaire measuring the frequency of complaints. Each item is scored 0-4 (0=never, 4=always). The final score is the sum of the scores of the 5 items (total score 0-20)
Pelvic Organ Prolapse | 11-13 weeks gestation
  Pelvic Organ Prolapse Distress Inventory
Pelvic Organ Prolapse | 28-33 weeks gestation
  Pelvic Organ Prolapse Distress Inventory
Pelvic Organ Prolapse | 3 months postpartum
  Pelvic Organ Prolapse Distress Inventory
Pelvic Organ Prolapse | 12 months postpartum
  Pelvic Organ Prolapse Distress Inventory
Sexual function | 11-13 weeks gestation
  POP/UI Sexual Questionnaire - IUGA revised
Sexual function | 28-33 weeks gestation
  POP/UI Sexual Questionnaire - IUGA revised
Sexual function | 3 months postpartum
  POP/UI Sexual Questionnaire - IUGA revised
Sexual function | 12 months postpartum
  POP/UI Sexual Questionnaire - IUGA revised

CONTACTS AND LOCATIONS:
Overall Officials: Jan Deprest, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lagaert L, Weyers S, Van Kerrebroeck H, Elaut E. Postpartum dyspareunia and sexual functioning: a prospective cohort study. Eur J Contracept Reprod Health Care. 2017 Jun;22(3):200-206. doi: 10.1080/13625187.2017.1315938. Epub 2017 Apr 27. PMID 28447919
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Result] Reimers C, Staer-Jensen J, Siafarikas F, Saltyte-Benth J, Bo K, Ellstrom Engh M. Change in pelvic organ support during pregnancy and the first year postpartum: a longitudinal study. BJOG. 2016 Apr;123(5):821-9. doi: 10.1111/1471-0528.13432. Epub 2015 Jun 26. PMID 26113145
- [Result] Skouteris H, Carr R, Wertheim EH, Paxton SJ, Duncombe D. A prospective study of factors that lead to body dissatisfaction during pregnancy. Body Image. 2005 Dec;2(4):347-61. doi: 10.1016/j.bodyim.2005.09.002. Epub 2005 Nov 21. PMID 18089200
- [Result] Clark A, Skouteris H, Wertheim EH, Paxton SJ, Milgrom J. The relationship between depression and body dissatisfaction across pregnancy and the postpartum: a prospective study. J Health Psychol. 2009 Jan;14(1):27-35. doi: 10.1177/1359105308097940. PMID 19129334
- [Result] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Result] Frank L, Kleinman L, Farup C, Taylor L, Miner P Jr. Psychometric validation of a constipation symptom assessment questionnaire. Scand J Gastroenterol. 1999 Sep;34(9):870-7. doi: 10.1080/003655299750025327. PMID 10522604
- [Result] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Result] Utomo E, Blok BF, Steensma AB, Korfage IJ. Validation of the Pelvic Floor Distress Inventory (PFDI-20) and Pelvic Floor Impact Questionnaire (PFIQ-7) in a Dutch population. Int Urogynecol J. 2014 Apr;25(4):531-44. doi: 10.1007/s00192-013-2263-z. Epub 2014 Jan 21. PMID 24445668
- [Result] Dietz HP. Pelvic floor ultrasound: a review. Am J Obstet Gynecol. 2010 Apr;202(4):321-34. doi: 10.1016/j.ajog.2009.08.018. PMID 20350640